CLINICAL TRIAL: NCT06250400
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled Parallel Study：Clinical Study of Efficacy and Safety of Histamine Human Immunoglobulin (ShuYangMinNing) in the Treatment of Chronic Spontaneous Urticaria (CSU)
Brief Title: Efficacy and Safety of Histamine Human Immunoglobulin in the Treatment of Chronic Spontaneous Urticaria (CSU)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hangzhou Grand Biologic Pharmaceutical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: I-23PJ2191
Record Dates: First submitted 2024-01-15; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — Loratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Treatment arm will receive a dose of Histamine Human Immunoglobulin 12mg (2ml) s.c. which consists of one injection of Histamine Human Immunoglobulin 12mg(2ml) vial every week for 4 times.
  Treatment arm will also receive a dose of loratadine p.o. which consists of one pill of loratadine 10mg every day for 4 weeks.
  Interventions: Biological: human histaglobulin; Drug: Loratadine 10 Mg
- Placebo (Placebo Comparator): Placebo arm will receive placebo which consists of one injection of placebo 12mg(2ml) vial every week for 4 times.
  Placebo arm will also receive a dose of loratadine p.o. which consists of one pill of loratadine 10mg every day for 4 weeks.
  Interventions: Biological: placebo; Drug: Loratadine 10 Mg

INTERVENTIONS:
Biological: human histaglobulin — once 12 mg/2ml/bottle, 2 subcutaneous injection once a week, using 4 times in a row, a total of 28 d;
  Arms: Treatment
Biological: placebo — once 12 mg/2ml/bottle, 2 subcutaneous injection once a week, using 4 times in a row, a total of 28 d;
  Arms: Placebo
Drug: Loratadine 10 Mg — orally, 10mg once a day for 4 weeks

SUMMARY:
The goal of this clinical trial is to study patients with chronic spontaneous urticaria. The main question it aims to answer is the efficacy and safety of histamine human immunoglobulin (ShuYangMinNing) in the treatment of chronic spontaneous urticaria.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed；
2. Age ≥ 18 years；
3. Meet the diagnostic criteria of chronic spontaneous urticaria from《Guideline for diagnosis and treatment of urticaria in China（2022）》and follow the doctor's advice；the patient had urticaria symptoms in the previous week before enrollment, and UAS7 score(range 0-42) ≥ 7;
4. Patients with uncontrolled urticaria are regularly treated with standard single-dose antihistamines regularly for 2 weeks before screening;

Exclusion Criteria:

1. Pregnant or nursing (lactating) women;
2. Patients with malignant tumors, severe liver and kidney diseases, hematological disorders, autoimmune diseases(such as systemic lupus erythematosus, Sjogren's syndrome, dermatomyositis, myositis, systemic vasculitis, systemic sclerosis, rheumatoid arthritis, spondyloarthropathy or other rheumatic immune diseases evaluated by the physician that are not suitable for inclusion), chronic serious infections, diabetic peripheral neuropathy, psychosis, and other diseases or medical histories that may affect normal efficacy evaluation and/or subject safety evaluation；
3. History of drug or alcohol abuse;
4. Patients who discontinue systemic use of glucocorticoids and other immunosuppressants(such as cyclosporin A, wilfordii , etc.) that affect immune function for less than 4 weeks;Patients who discontinue systemic use of biologics (e.g., omalizumab) for less than 3 months;
5. Patients with symptoms of urticaria and/or angioedema, Including but not limited to urticaria vasculitis, serum sickness like reaction, bullous pemphigoid, mastocytosis, neutrophilic urticaria dermatosis, Schnitzler syndrome, autoinflammatory response syndromes (e.g., tumor necrosis factor receptor-associated periodic fever syndrome, familial Mediterranean fever, mevaldate kinase deficiency, etc.);or other chronic itchy skin conditions, such as atopic dermatitis, dermatitis herpetiformis, and pruritus senile;
6. Allergic to human immunoglobulin;
7. History of other severe allergic reactions;
8. Patients with pathological arrhythmias and a history of organic heart disease; Patients with known or suspected QT prolongation; or patients who are unable to discontinue medications that cause QT prolongation during the trial；
9. Subjects whom the investigator considers unsuitable for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2024-03-31 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease control rate during the last week of treatment (i.e., proportion of patients with urticaria activity score for 7d（UAS7，range 0-42) < 7 for 7 consecutive days after the last injection) | through study completion, an average of 1 year
  The Urticaria Activity Score (UAS) is a composite, diary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for the number of wheals (hives) and the intensity of the pruritus (itch) . The daily UAS is calculated as the average of the morning and evening scores. The urticaria activity score for 7d (UAS7) is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. UAS7 scores ranged from 0 to 42. If UAS7 score is less than 7, it indicates disease control.
  A minimum of 4 out of 7 daily scores were needed to calculate the UAS7 values. Otherwise, the weekly score was missing for that week.
  The primary outcome measure was disease control rate in the last week of treatment. Chi-square test was used for comparison between groups. Based on the analysis for the main full analysis set (FAS), based on the analysis of the per protocol set（PPS) for supporting analysis.

SECONDARY OUTCOMES:
Time when UAS7 (range 0-42) <7 for the first time | up to 5 weeks
  The Urticaria Activity Score (UAS) is a composite, diary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for the number of wheals (hives) and the intensity of the pruritus (itch) . The daily UAS is calculated as the average of the morning and evening scores. The UAS7 is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. UAS7 scores ranged from 0 to 42. A higher UAS7 indicated greater urticaria disease activity.If UAS7 score is less than 7, it indicates disease control.
Changes in UAS7 scores(range 0-42) after each dose compared with baseline | up to 5 weeks
  The Urticaria Activity Score (UAS) is a composite, diary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for the number of wheals (hives) and the intensity of the pruritus (itch) . The daily UAS is calculated as the average of the morning and evening scores. The UAS7 is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. UAS7 scores ranged from 0 to 42. A higher UAS7 indicated greater urticaria disease activity.If UAS7 score is less than 7, it indicates disease control.
Proportion of patients who responded to treatment as assessed by UCT score | up to 5 weeks
  The urticaria control test (UCT) is a recently validated tool for disease control assessment in patients with CSU.Disease control over the past 4 weeks was evaluated retrospectively. The assessment included: ①the occurrence of urticaria symptoms (such as itching, wheals, etc.); ②the impact of quality of life; ③the frequency of symptoms was not sufficiently controlled by the treatment; ④overall disease control status. The score of each item ranged from 0 to 4, and the total score was the sum of the scores of the four questions.A score of 0 indicates that the disease is not under control at all, and a score of 16 indicates that it is under complete control. A total score ≥12 indicated well-controlled urticaria, and a score < 12 indicated poorly controlled urticaria.When UCT increased by ≥ 3 points, the current treatment regimen was effective.
Proportion of patients with well-controlled disease as assessed by UCT score | up to 5 weeks
  The urticaria control test (UCT) is a recently validated tool for disease control assessment in patients with CSU.Disease control over the past 4 weeks was evaluated retrospectively. The assessment included: ① the occurrence of urticaria symptoms (such as itching, wheals, etc.); ② the impact of quality of life; ③ the frequency of symptoms was not sufficiently controlled by the treatment; ④ overall disease control status. The score of each item ranged from 0 to 4, and the total score was the sum of the scores of the four questions.A score of 0 indicates that the disease is not under control at all, and a score of 16 indicates that it is under complete control. A total score ≥12 indicated well-controlled urticaria, and a score < 12 indicated poorly controlled urticaria.When UCT increased by ≥ 3 points, the current treatment regimen was effective.
Change in chronic urticaria quality of life questionnaire (CU-Q2oL) score from baseline | up to 5 weeks
  The Chronic Urticaria Quality of Life Questionnaire(CU-Q2oL) contains 23 items to assess the impairment of health-related quality of life (HR-QOL) in the past 2 weeks from pruritus, swelling, effect on daily activities, sleep problems, limitation and appearance. The scores of 23 items were added and linearly transformed to a total score of 0-100 CU⁃Q2oL can not only use the total score of the questionnaire to represent the overall damage of HR⁃QoL, but also use the score of one aspect (dimension) to represent the damage of specific HR⁃QoL. The higher the score, the more severe the impact of CSU on the patient.
Proportion of patients who developed respiratory infections | up to 10 weeks
  Assess the proportion of patients who developed respiratory infections during the study

OTHER OUTCOMES:
Dosage of loratadine tablets and ebastine tablets | up to 10 weeks
  Assess the dosage of loratadine tablets and ebastine tablets
The Amount of Histamine, autoantibodies and FcepsilonRI receptors | up to 10 weeks
  Assess the Histamine, autoantibodies, and immunoglobulin E binds to the high-affinity Fcepsilon receptor I (FcepsilonRI) receptors

IPD SHARING:
Plan to Share IPD: No